CLINICAL TRIAL: NCT05727280
Title: The Effect of Progressive Relaxation Exercise on Pain Level, Sleep Quality and Analgesic Consumption of Patients Undergoing Open Heart Surgery: a Randomized Controlled Study
Brief Title: The Effect of Progressive Relaxation Exercise on Pain Level, Sleep Quality and Analgesic Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Gamze Bolattürk, Research Assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GBolatturk
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pain Level, Sleep Quality and Analgesic Consumption in Open Heart Surgery
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled single-blind quasi-experimental research design.
Who Masked: Participant
Masking Description: In the randomization process, those who meet the criteria for inclusion in the sample and accept to participate in the study do not know that they will be included in the intervention group or the control group, so it will be single-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): After the first meeting with the patients in the intervention group, the patients will be informed about the application of the Progressive Relaxation Exercise and the exercise application will be taught. After open heart surgery, progressive relaxation exercise will be applied to the patient on the 1st, 2nd and 3rd days of his admission to the service. The patient will be asked to perform the progressive relaxation exercise twice a day, once during the day and once in the evening. Before each daytime application, the score given by the patient to the SF-MPQ will be recorded. Patients will be asked to repeat the same application two hours after dinner. In the morning of the next day after each application, the score given by the patient to the RCSQ will be recorded by the researcher.
  Interventions: Behavioral: Progressive Relaxation Exercise Practices
- Control Group (No Intervention): After the first meeting with the patients in the control group, the routine care and treatment practices planned by the service will continue. No additional intervention is planned for the patients in this group. After open heart surgery, patients will be asked to fill out the SF-MPQ and RCSQ on the 1st, 2nd and 3rd days of the patient's admission to the service. After the completion of the study, progressive relaxation exercise training will be given to the patients in the control group.

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercise Practices — The intervention planned within the scope of the research are the Progressive Relaxation Exercise application. Patients in the intervention group undergoing open heart surgery will be given training on progressive relaxation exercise in the patient's room the day before the surgery. Correct breathing techniques will be taught and the relaxation exercises will be performed by using audio recordings. Afterwards, the relaxation exercise will be provided to the patient to practice the progressive relaxation exercise with mp3 accompaniment. After open heart surgery, progressive relaxation exercise will be applied to the patient on the 1st, 2nd and 3rd days of his admission to the service. The patient will be asked to perform the progressive relaxation exercise twice a day, once during the day and once in the evening.
  Arms: Intervention Group

SUMMARY:
Coronary artery bypass graft (CABG) surgery is the process of providing re-oxygenation of the myocardium by anastomosis to the occluded heart coronary with the graft created using certain vessels of the body. After CABG surgery, pain occurs due to thoracic surgical incision, surgical incision in the saphenous vein or radial artery regions for grafting. Pain that is not well managed in the post-operative period also increases the analgesic consumption of the patients. When pain management is inadequate, the patient's recovery process is affected by causing limitation in movements, digestive, circulatory, respiratory system and sleep problems in the postoperative period.

Progressive relaxation exercise (PRE) is an application that provides relaxation and relaxation as a result of conscious contraction and relaxation of large muscle groups in the body, and increasing body awareness in the individual. PRE is among the preferred non-pharmacological applications today in terms of being inexpensive, harmless, easily administered by the patient, positively affecting the patient's functions and reducing their complaints. Studies have generally evaluated the effectiveness of pharmacological (analgesic) methods in order to reduce postoperative pain. Although analgesics are indispensable in the management of postoperative pain, they may not always be sufficient to reduce the patient's pain sufficiently. Also, analgesics have some undesirable side effects. For this reason, it is reported that the use of non-pharmacological methods together with pharmacological methods increases the effectiveness of pharmacological methods in order to reduce the pain experienced by the patients after the surgical intervention and to reduce the complaints that occur in the patient due to pain. For this reason, various analgesic combinations and non-pharmacological methods should be used together to reduce postoperative pain. In this direction, PRE has become a technique frequently used and preferred by nurses in pain management in recent years.

The PGE technique, developed by Jacobson in 1929, is based on the idea that anxiety-provoking thoughts and events create physiological tension. PGE is the conscious contraction and relaxation of large muscle groups in the body, and noticing the change in between. PGE can be performed one-on-one or as a group in one or several sessions with the help of a CD or audio recorder. It can be applied with musical accompaniment, visual imagery or diaphragmatic breathing to increase its effectiveness. The exercise can be done from head to foot or from foot to head. In this study, it was aimed to investigate the effect of progressive relaxation exercise on postoperative pain level, sleep quality and analgesic consumption in patients undergoing open heart surgery.

DETAILED DESCRIPTION:
One of the non-pharmacological treatment methods that can provide therapeutic benefit for pain management and improving sleep quality is Progressive relaxation exercise (PRE). The PRE is the conscious contraction and relaxation of large muscle groups in the body, and noticing the change (Demir Burcu, 2013; Genç and Oğuz, 2018; Oğuz et al., 2019). The PRE technique, developed by Jacobson in 1929, is based on the idea that anxiety-provoking thoughts and events create physiological tension (Blanaru, 2012). Jacobson developed the PRE to raise awareness of skeletal muscle tension. Muscle tension is triggered by various negative emotions and psychosomatic diseases. With this exercise, relaxation is aimed to reduce the feeling of tension and the perceived stress level (Genç & Oğuz, 2018; Oğuz et al., 2019). The PRE; it is an inexpensive method that can be easily taught by nurses, yoga instructors, clinical psychologists, and other complementary alternative medicine practitioners. The PRE can be performed one-on-one or as a group in one or several sessions with the help of a CD or audio recorder. It can be applied with musical accompaniment, visual imagery or diaphragmatic breathing in order to increase its effectiveness (Genç and Oğuz, 2018; Oğuz et al., 2019). The PRE involves sequentially stretching and relaxing all 16 muscle groups as you breathe in. The exercise can be from head to foot or from foot to head. During the exercise, the patient must complete the processes of perceiving the tension in his body, maintaining control and being able to go into a state of relaxation. After the patient is informed about the exercise, he starts with breathing exercises. A deep but relaxing breath is taken through the nose, and simultaneously with the relaxation, the lips are contracted and breath given through the mouth. During this application, the patient keeps the muscle group he is working in for 10 seconds; the nurse, on the other hand, enables the patient to notice the warmth/warming felt in the muscle group (Demiralp, 2006; Demiralp & Oflaz, 2007; Ratfisch, 2015; Demiralp & Oflaz, 2011; Özveren, 2011; Eyüpoğlu, 2013). In order for PRE to be effective, there must be no factors that can warn the patient, and the room must be dim, airy and at a suitable temperature. During the exercise, the patient is asked to sit in a comfortable chair or lie on his back. Effective work does not occur because it is loaded on some muscle groups in the side or prone position. The patient should be physically and mentally comfortable. In order to achieve this, the clothes should be chosen loosely and there should be no items (belt, buckle, glasses, etc.) that will tighten the body. In the mental sense; It should be ensured that he can focus on a tool (sound, word, object, etc.) in order to get away from the bad thoughts in his mind (Yıldırım, 1991; McCallie et al., 2006; Özveren, 2011).

In this study, it is aimed to evaluate the effect of progressive relaxation exercise applied to patients undergoing cardiac surgery on pain level, sleep quality and analgesic consumption. In addition, it is thought that the results obtained from this study will increase awareness of progressive relaxation exercise and other similar applications as a cheap, easy, effective, applicable and easily adaptable non-pharmacological method in patients undergoing cardiac surgery. The research hypotheses are:

1. Progressive relaxation exercise have an effect on pain level in patients undergoing open heart surgery.
2. Progressive relaxation exercise have an effect on sleep quality in patients undergoing open heart surgery.
3. Progressive relaxation exercise have an effect on analgesic consumption in patients undergoing open heart surgery.
4. There is a difference between the pain level, sleep quality and analgesic consumption of the patients who underwent open heart surgery in the intervention group, in which progressive relaxation exercise was applied, and in the control group, which was not applied progressive relaxation exercise.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone open heart surgery and heart valve surgery
* Being extubated within the first 4 hours after CABG and heart valve surgery
* Being transfer to service within 48-72 hours after CABG and heart valve surgery
* Being between 30 and 85 years old
* Having ability to read, write and speak Turkish
* Being conscious and oriented
* Having no problems communication
* Not experiencing any psychological discomfort
* Having no problems with seeing, hearing, speaking and expressing oneself
* No complications before, during and three days after surgery
* Beeing volunteer and agree to participate in research

Exclusion Criteria:

* Having a speech and hearing problem that prevents the understanding of the given information and the application of PRE
* Presence of diagnosed neurological or psychiatric disease
* Being a foreign national
* Being unconscious in the pre- and postoperative period

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Critical-Care Pain Observation Tool (CPOT) | within 48-72 hours of patients staying in intensive care
  Critical-Care Pain Observation Tool (CPOT) will be used to determine the pain intensity of the participants in the intensive care unit. The CPOT Gèlinas et al. was developed by at 2007. The Turkish validity and reliability study of the scale was performed by Gündoğan et al. made by at 2016. The scale includes four subscales, including facial expression, muscle tension, body movements, and compliance with ventilation in intubated patients, and behavioral items consisting of sounds made in extubated patients. Each of the subscales of the scale is evaluated between 0-2 points and the total score of the scale varies between 0-8. The intensive care pain observation scale can be used both in patients who can communicate verbally and in intubated and deep sedation situation. The CPOT is a valid and reliable scale to evaluate the pain of intensive care patients. Scores above 2 in the CPOT indicate that the patient is experiencing pain.

SECONDARY OUTCOMES:
Short Form McGill Pain Questionnaire (SF-MPQ) | The 1st, 2nd and 3rd days of the patient's in the service after open heart surgery
  Short Form McGill Pain Questionnaire (SF-MPQ), which was developed by Melzack in 1987, provides information about the sensory characteristics of the pain, the severity of pain and its effects. Its validity and reliability in our country Yakut et al. by performed at 2007. It includes three different sections within the SF-MPQ.
  First Part (pain form): This part includes words that give information about the nature of the pain felt. In this part of the scale, a total of three pain scores are obtained: sensory pain score, perceptual pain score and total pain score.
  Second Part (current pain index): This part includes five different word groups that can range from "mild pain" to "unbearable pain" to determine the severity of the pain described by the patient.
  Third Part (pain scale score): Individuals are asked to mark on a 10 cm long scale in the visual analog part of the pain intensity, taking into account the current severity of the pain felt.
Richard-Campbell Sleep Questionnaire (RCSQ) | The 1st, 2nd and 3rd days of the patient's in the service after open heart surgery
  Richard-Campbell Sleep Questionnaire (RCSQ) was developed in 1987 to describe sleep problems experienced at night. The scale consists of 6 questions that measure the characteristics of the previous night's sleep (depth of night sleep, time to fall asleep, frequency of awakening, time to stay awake when awakened, sleep quality and noise level in the environment). The first 5 questions are included in the scale scoring, and the 6th question is excluded from the scoring. Each item in the scale is evaluated on a scale between 0 and 100, increasing with 5-point intervals (0-5-10-15-.....-90-95-100). If the scores obtained from the scale are between "0-25", it indicates very poor sleep quality, and between "76-100" indicates very good sleep quality. The higher the score, the higher the sleep quality. The validity and reliability of the scale in our country; It was made by Özlü and Özer at 2015.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Bolattürk, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University Hospital, Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No